CLINICAL TRIAL: NCT03805360
Title: The Erector Spinae Plane Block and Its Effect on Respiratory Status and Pain Management in Rib Fracture Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20014264
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Ropivacaine; Anesthetics, Local; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study aims to assess the systemic absorption of ropivacaine when it is administered into the erector spinae plane compartment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESP block with normal saline (Sham Comparator): An erector spinae plane block will be performed and a single dose of Normal Saline Flush, 0.9% Injectable Solution will be administered into the target muscle plane.
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution
- ESP block with local anesthetic (Experimental): An erector spinae plane block will be performed and a single dose of 0.5% ropivacaine will be injected into the target muscle plane.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine is a local anesthetic that is expected to provide numbness to the chest wall when injected into the erector spinae plane.
  Other Names: Local anesthetic
  Arms: ESP block with local anesthetic
Drug: Normal Saline Flush, 0.9% Injectable Solution — Normal Saline Flush, 0.9% Injectable Solution is not expected to provide numbness to the chest wall when injected into the erector spinae plane.
  Other Names: 0.9% Sodium Chloride
  Arms: ESP block with normal saline

SUMMARY:
The purpose of this research study is to identify the benefits of a type of nerve block, called an erector spinae plane block (ESP), in the treatment of patients with multiple rib fractures and uncontrolled pain despite receiving current institutional standards of care.

DETAILED DESCRIPTION:
Rib fractures are one of the most common injuries secondary to blunt chest trauma, and carry significant risk in terms of patient morbidity and mortality. Pulmonary complications resulting from these injuries include severe atelectasis with hypoxemia, pneumonia, pleural effusions, respiratory distress syndrome, need for mechanical ventilation and ICU admission, and prolonged hospital stay. Many institutions have tried to develop protocols to risk stratify and appropriately treat these patients, with the goal of predicting those with higher likelihood of pulmonary complications in order to minimize additional morbidity. Studies have demonstrated critical spirometry values which correlate to worse patient outcomes; specifically, vital capacity less than 50% predicted, or less than 2L. Subsequently, there have been numerous attempts to identify the best treatment interventions for these high risk patients. In addition to multi-modal pain management, the most commonly used procedures include thoracic epidurals, continuous or single shot paravertebral blocks, and intercostal blocks. However, all of the above interventions carry significant risk, and the frequent use lovenox thromboprophylaxis drastically limit their use. Recently, a novel peripheral nerve block technique has been developed, an erector spinae plane block (ESP), which may provide similar or greater efficacy to the above, with significantly less risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Blunt chest trauma
* Sustaining at least 3 unliateral rib fractures
* Resultant vital capacity less than 30% predicted
* Pain score reaches threshold despite using the current institutional standard of care for pain control

Exclusion Criteria:

* Patients whose weight less than 60kg.
* Patients with bilateral rib fractures.
* Patients that are intubated and mechanically ventilated.
* Pregnant Individuals.
* Any individual with a documented allergy to ropivacaine.
* Patients with limited English proficiency (LEP)
* Patients whose body habitus prevents the practitioner's ability to adequately perform the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change in numeric pain score rating at rest (before incentive spirometry exercise) | Baseline and at 45 minutes after ESP block
  Self-reported pain intensity before the ESP block is performed and after the ESP block is performed. These measurements will be assessed before the incentive spirometry exercise. Each item is scored 0-10 (0 = no pain; 10= worst pain possible)
Change in numeric pain score rating with respiration (after incentive spirometry exercise) | Baseline and at 45 minutes after ESP block
  Self-reported pain intensity before the ESP block is performed and after the ESP block is performed. These measurements will be assessed after the incentive spirometry exercise. Each item is scored 0-10 (0 = no pain; 10 = worst pain possible)
Change in incentive spirometry values | Baseline and at 45 minutes after ESP block
  Incentive spirometry values, measured in cubic centimeters, when the participant provides one inhalational breath at maximum effort. The first measurement will be taken before the ESP block procedure and the second measurement 45 minutes after the ESP block procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Tran, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03805360/Prot_SAP_000.pdf